CLINICAL TRIAL: NCT00856830
Title: Phase I/IIa Study of the Novel Combination of Bendamustine With Irinotecan Followed by Etoposide/Carboplatin in Chemonaive Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Bendamustine With Irinotecan Followed by Etoposide/Carboplatin for Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Francisco Robert,MD, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F080929010; UAB 0818 (Other: Institutional study protocol number)
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Small Cell Lung Cancer; Extensive Stage Lung Cancer; Chemonaive
Keywords: Small cell lung cancer; Chemonaive; Bendamustine; Irinotecan; Etoposide; Carboplatin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Carboplatin; Etoposide; Bendamustine Hydrochloride

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label, Phase I - II trial with an initial dose escalation component and an expansion cohort of patients treated at the recommended Phase II dose.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Novel Drug Combination (Experimental): This novel drug combination includes: Bendamustine, Irinotecan, and Etoposide/Carboplatin.
  This study has only one arm but it incorporates two phases. Phase I utilizes a combination of bendamustine and irinotecan for Regimen A followed by etoposide and carboplatin for Regimen B.
  Interventions: Drug: Novel Drug Combination

INTERVENTIONS:
Drug: Novel Drug Combination — This novel drug combination includes: Bendamustine, Irinotecan, and Etoposide/Carboplatin. Subjects will be treated with irinotecan (150 mg/m2) infusion on Day 1 followed by infusion of bendamustine on Days 1 and 2 at increasing dose levels using a 3+3 design (starting dose of 80-mg/m2/d with 20 mg/mg/d incremental increase to max 120 mg/m2/d) (Regimen A). This will be repeated every 3 weeks for a total of 3 cycles. Restaging for response will be performed prior to the next regimen.
  * All subjects will then be given carboplatin (AUC 6) on day 1 and etoposide (100 mg/m2) on days 1, 2 and 3 (Regimen B). They will receive 3 cycles of this regimen every 3 weeks prior to restaging.
  * At the end (3 weeks after) of the sixth total round of chemotherapy, subjects will be re-evaluated for response, and will be followed-up for recurrent disease every 8 weeks.
  Other Names: Irinotecan (Camptosar); Carboplatin (Paraplatin); Etoposide (VdPesid); Bendamustine (Treanda)

SUMMARY:
Small cell lung cancer, or SCLC, constitutes approximately 15% of the 170,000 new cases of lung cancer diagnosed annually in the United States. Extensive-stage SCLC comprises two thirds of new cases and is generally considered sensitive to chemotherapy, despite a median time to progression of 4 months. SCLC is one of the most aggressive and lethal types of cancer, with a median survival of 9 months (range 7-11 months) in patients diagnosed with extensive disease. Overall, the majority of patients with SCLC die in less than 2 years (2-year survival rates generally less than 10%), and the 5-year survival rate is 2.3% for patients with extensive disease. The regimen of etoposide in combination with a platinum (cisplatin or carboplatin) is generally considered the "standard of care" although a recent Phase III trial suggests improved survival with the combination of cisplatin/irinotecan. Further evaluation of new agents in combination regimens attempting to overcome the intrinsic drug resistance seen in extensive-stage SCLC is warranted attempting to improve survival and achieve palliation of disease-related symptoms.

DETAILED DESCRIPTION:
We are proposing a novel combination of bendamustine plus irinotecan followed by the standard regimen of etoposide with carboplatin. This will allow the investigation of response to the novel combination as well as any improvement in outcomes compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of extensive stage SCLC.
* Measurable or assessable tumor parameters.
* ECOG Performance Status 0-2.
* Age between 18 and 79 years (in the State of Alabama > 18).
* Adequate bone marrow, liver and renal function, defined as:
* Absolute neutrophil count (ANC) ≥ 1500/µL
* Hemoglobin ≥ 8g/dl
* Platelet count ≥ 100,000/µL
* SGOT/SGPT ≤ 2 x upper limit of normal or ≤ 5 x upper limit of normal when liver metastases are present.
* Total bilirubin value ≤ 2 x upper limit of normal.
* Serum creatinine value ≤ 2 x upper limit of normal.
* Fully recovered from any previous surgery (at least 4 weeks since major surgery)
* Must have recovered from prior radiation therapy (at least 3 weeks)
* All subjects must agree to practice approved methods of birth control (if applicable). A negative pregnancy test must be documented during the screening period for women of childbearing potential.
* Must provide written informed consent and authorization to use and disclose health information (HIPAA).
* Extensive-stage SCLC as defined as disease not confined to one hemithorax, including ipsilateral pleural effusion or pericardial effusion.
* No prior chemotherapy.

Exclusion Criteria:

* Concurrent cancer chemotherapy, biologic therapy or radiotherapy.
* Administration of any investigational drug within 28 days prior to administration of the current therapy.
* Symptomatic brain metastases; those patients should be treated first with either whole brain radiation therapy or radiosurgery.
* Concurrent serious infection.
* Concomitant severe or uncontrolled underlying medical disease unrelated to the tumor, which is likely to compromise patient safety and affect the outcome of the study.
* History of other malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for a minimum of 2 years.
* Neuropathy at baseline ≥ Grade 2.
* Any evidence or history of hypersensitivity or other contraindications for the drugs used in this trial.
* History of chronic diarrhea; or diarrhea (excess of 2-3 stools/day above normal frequency) in the past 2 weeks.
* History of a positive serology for human immunodeficiency virus (HIV).
* Psychiatric disorder that prevents patients from providing informed consent or following protocol instructions.
* Pregnant or lactating women.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Georgia Cancer Specialists, Marietta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: April 2009, Primary Completion Date: May 2015 and Study Completion Date: May 2016. Recruitment location: University of Alabama at Birmingham and Georgia Cancer Specialists.
Pre-assignment Details: We are proposing a novel combination of bendamustine plus irinotecan followed by the standard regimen of etoposide with carboplatin. This will allow the investigation of response to the novel combination as well as any improvement in outcomes compared to historical controls.
Groups:
- Phase I - Regimen A: Cohort I (80 mg/m2) - Bendamustine (B): Participants were treated with irinotecan at 150 mg/m2 on day 1 followed by bendamustine (80 mg/m2) on days 1 and 2: every 21 days for a total of 3 cycles Participants with either objective response or stable disease after 3 cycles of Regimen A, received Regimen B as a consolidation. Carboplatin AUC6 (Day 1), Etoposide 100mg/m2 (Day 1,2,3) every 21 days for 3 cycles.
- Phase I - Regimen A: Cohort II 100mg/m2) - (B): Participants were treated with irinotecan at 150 mg/m2 on day 1 followed by bendamustine (100 mg/m2) on days 1 and 2: every 21 days for a total of 3 cycles.
  Participants with either objective response or stable disease after 3 cycles of Regimen A, received Regimen B as a consolidation. Carboplatin AUC6 (Day 1), Etoposide 100mg/m2 (Day 1,2,3) every 21 days for 3 cycles.
- Phase I - Regimen A: Cohort III (120 mg/M2) - (B): Participants were treated with irinotecan at 150 mg/m2 on day 1 followed by bendamustine (120 mg/m2) on days 1 and 2: every 21 days for a total of 3 cycles.
  Participants with either objective response or stable disease after 3 cycles of Regimen A, received Regimen B as a consolidation. Carboplatin AUC6 (Day 1), Etoposide 100mg/m2 (Day 1,2,3) every 21 days for 3 cycles.
- Phase II - Regimen A: Cohort IV (B) 100 -120 mg/m2 (Day 1,2): Participants were treated with irinotecan at 150 mg/m2 on day 1 followed by bendmustine on days 1 and 2 at bendamustine 100-120 mg/m2 (Day 1,2). This was repeated every 21 days for a total of 3 cycles.
  Participants with either objective response or stable disease after 3 cycles of Regimen A, received Regimen B as a consolidation. Carboplatin AUC6 (Day 1), Etoposide 100mg/m2 (Day 1,2,3) every 21 days for 3 cycles.
Period: Irinotecan & Bendamustine
Arm/Group | Phase I - Regimen A: Cohort I (80 mg/m2) - Bendamustine (B) | Phase I - Regimen A: Cohort II 100mg/m2) - (B) | Phase I - Regimen A: Cohort III (120 mg/M2) - (B) | Phase II - Regimen A: Cohort IV (B) 100 -120 mg/m2 (Day 1,2)
Started | 3 | 6 | 6 | 15
Maximum Tolerated Dose | 3 | 6 | 6 | 12
Completed | 3 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1
Period: Regimen - B (Carboplatin & Etoposide)
Arm/Group | Phase I - Regimen A: Cohort I (80 mg/m2) - Bendamustine (B) | Phase I - Regimen A: Cohort II 100mg/m2) - (B) | Phase I - Regimen A: Cohort III (120 mg/M2) - (B) | Phase II - Regimen A: Cohort IV (B) 100 -120 mg/m2 (Day 1,2)
Started | 3 | 6 | 6 | 12
Completed | 3 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Regimen A: Cohort I Bendamustine 80 mg/m2 (Day 1,2): Participants were treated with irinotecan at 150 mg/m2 on day 1 followed by bendmustine on days 1 and 2 at increasing dose levels using a 3 + 3 design. The initial dose of bendamustine was 80 mg/m2 with incremental 20 mg/m2 dose escalation to a maximum of 120 mg/m2. This was repeated every 21 days for a total of 3 cycles.
- Regimen A: Cohort II Bendamustine 100 mg/m2 (Day 1,2): Participants were treated with irinotecan at 150 mg/m2 on day 1 followed by bendmustine on days 1 and 2 at increasing dose levels using a 3 + 3 design. The initial dose of bendamustine was 100 mg/m2 with incremental 20 mg/m2 dose escalation to a maximum of 120 mg/m2. This was repeated every 21 days for a total of 3 cycles.
- Regimen A: Cohort III Bendamustine 120 mg/m2 (Day 1,2): Participants were treated with irinotecan at 150 mg/m2 on day 1 followed by bendmustine on days 1 and 2 at increasing dose levels using a 3 + 3 design. The initial dose of bendamustine was 120 mg/m2 with incremental 20 mg/m2 dose escalation to a maximum of 120 mg/m2. This was repeated every 21 days for a total of 3 cycles.
- Regimen A: Cohort IV Bendamustine 100 -120 mg/m2 (Day 1,2): Participants were treated with irinotecan at 150 mg/m2 on day 1 followed by bendmustine on days 1 and 2 at increasing dose levels using a 3 + 3 design. Bendamustine was given at 100 - 120 mg/m2. This was repeated every 21 days for a total of 3 cycles.
- Total: Total of all reporting groups
Arm/Group | Regimen A: Cohort I Bendamustine 80 mg/m2 (Day 1,2) | Regimen A: Cohort II Bendamustine 100 mg/m2 (Day 1,2) | Regimen A: Cohort III Bendamustine 120 mg/m2 (Day 1,2) | Regimen A: Cohort IV Bendamustine 100 -120 mg/m2 (Day 1,2) | Total
Number analyzed (Participants) | 3 | 6 | 6 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 5 | 13 | 27
  >=65 years | 0 | 0 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7 | 14
  Male | 1 | 3 | 4 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 6 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicity Regimen A - Phase I
Description: The determination of the dose limiting toxicity as defined by The National Cancer Institute Common Toxicity Criteria version 3 as follows: grade 4 neutropenia >5 days; grade 3/4 febrile neutropenia; grade 4 thrombocytopenia; or grade >2 non-hematologic toxicities (except for nausea/vomiting, alopecia, or fatigue).
Time Frame: 9 weeks
Measure: Number; unit: participants
Groups:
- Novel Drug Combination: There is only one arm but it incorporates two phases. Phase I utilizes a combination of bendamustine and irinotecan for Regimen A followed by etoposide and carboplatin for Regimen B.
  Bendamustine, Irinotecan, Etoposide/Carboplatin (Novel drug combination): Subjects will be treated with irinotecan (150 mg/m2) infusion on Day 1 followed by infusion of bendamustine on Days 1 and 2 at increasing dose levels using a 3+3 design (starting dose of 80-mg/m2/d with 20 mg/mg/d incremental increase to max 120 mg/m2/d) (Regimen A). This will be repeated every 3 weeks for a total of 3 cycles. Restaging for response will be performed prior to the next regimen.
  * All subjects will then be given carboplatin (AUC 6) on day 1 and etoposide (100 mg/m2) on days 1, 2 and 3 (Regimen B). They will receive 3 cycles of this regimen every 3 weeks prior to restaging.
  * At the end (3 weeks after) of the sixth total round of chemotherapy, subjects will be re-evaluated for response, and will be followed
Arm/Group | Novel Drug Combination
Number analyzed (Participants) | 15
participants
  Phase I - Cohort I | 0
  Phase I - Cohort II | 1
  Phase I - Cohort III | 1

2. Primary Outcome: Number of Patients With Adverse Events - Phase II
Description: The degree of toxicity as defined by The National Cancer Institute Common Toxicity Criteria version 3.
Time Frame: 9 weeks
Measure: Number; unit: participants
Groups:
- Novel Drug Combination: This novel drug combination includes: Bendamustine, Irinotecan, and Etoposide/Carboplatin.
  This study has only one arm but it incorporates two phases. Phase I utilizes a combination of bendamustine and irinotecan for Regimen A followed by etoposide and carboplatin for Regimen B.
  Novel Drug Combination: This novel drug combination includes: Bendamustine, Irinotecan, and Etoposide/Carboplatin. Subjects will be treated with irinotecan (150 mg/m2) infusion on Day 1 followed by infusion of bendamustine on Days 1 and 2 at increasing dose levels using a 3+3 design (starting dose of 80-mg/m2/d with 20 mg/mg/d incremental increase to max 120 mg/m2/d) (Regimen A). This will be repeated every 3 weeks for a total of 3 cycles. Restaging for response will be performed prior to the next regimen.
  •All subjects will then be given carboplatin (AUC 6) on day 1 and etoposide (100 mg/m2) on days 1, 2 and 3 (Regimen B). They will receive 3 cycles of this regimen every 3 weeks prior to restaging.
Arm/Group | Novel Drug Combination
Number analyzed (Participants) | 15
participants | 8

3. Secondary Outcome: Progression Free Survival
Description: Using the Response Evaluation Criteria in Solid Tumors (RECIST 2000), progression is defined as 20% or greater increase from the baseline tumor parameters or new lesions.
Time Frame: 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Novel Drug Combination
Number analyzed (Participants) | 27
months | 6.0 [4.0 to 7.0]

ADVERSE EVENTS:
Time Frame: 9 Weeks
Groups:
- Novel Drug Combination: This novel drug combination includes: Bendamustine, Irinotecan, and Etoposide/Carboplatin.This study has only one arm but it incorporates two phases. Phase I utilizes a combination of bendamustine and irinotecan for Regimen A followed by etoposide and carboplatin for Regimen B.
  Novel Drug Combination: This novel drug combination includes: Bendamustine, Irinotecan, and Etoposide/Carboplatin. Subjects will be treated with irinotecan (150 mg/m2) infusion on Day 1 followed by infusion of bendamustine on Days 1 and 2 at increasing dose levels using a 3+3 design (starting dose of 80-mg/m2/d with 20 mg/mg/d incremental increase to max 120 mg/m2/d) (Regimen A). This will be repeated every 3 weeks for a total of 3 cycles. Restaging for response will be performed prior to the next regimen.
  •All subjects will then be given carboplatin (AUC 6) on day 1 and etoposide (100 mg/m2) on days 1, 2 and 3 (Regimen B). They will receive 3 cycles of this regimen every 3 weeks prior to restaging.
Arm/Group | Novel Drug Combination
All-Cause Mortality (participants affected / at risk) | 2/30
Serious Adverse Events (participants affected / at risk) | 15/30
Other Adverse Events (participants affected / at risk) | 15/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novel Drug Combination (N=30)
Neutropenia (Blood and lymphatic system disorders) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 15 (15)
Fatigue (General disorders) | 10 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novel Drug Combination (N=30)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Nausea & Vomiting (Gastrointestinal disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Fatigue (General disorders) | 15 (15)
Neuropathy (Nervous system disorders) | 3 (3)
HyperKalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No